CLINICAL TRIAL: NCT01966263
Title: Fast-track Rehabilitation Protocol for Total Knee Arthroplasty: A Randomized Controlled Trial Comparing Local Infiltration Analgesia With Femoral Nerve Block
Brief Title: Fast Track Total Knee Arthroplasty: Local Infiltration Analgesia vs Femoral Nerve Block
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sint Maartenskliniek (Other)
Responsible Party: Principal Investigator, Maaike Fenten, Anesthesiologist, Head of anesthesiology department, Sint Maartenskliniek
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 497; 2013-001008-13 (EudraCT Number); NL43965.072.13 (Other: CCMO register)
Record Dates: First submitted 2013-10-11; First posted 2013-10-21 (Estimated); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-04

CONDITIONS: Arthroplasty, Replacement, Knee
Keywords: total knee arthroplasty; femoral nerve block; local infiltration analgesia; fast track
MeSH Terms: interventions — Epinephrine; Catheters; Saline Solution

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Infiltration Analgesia (LIA) (Active Comparator): local infiltration analgesia is an anesthetic technique that consists of the infiltration of operated tissue with a long acting local anesthetic during surgery to achieve postoperative pain relieve. In this study LIA of the knee will exist of: 1. local infiltration analgesia (LIA) of the posterior capsule of the knee, 2. LIA of the anterior capsule of the knee and 3. LIA of the subcutaneous tissue of the knee
  Interventions: Procedure: LIA of the posterior capsule of the knee; Procedure: LIA of the anterior capsule of the knee; Procedure: LIA of the subcutaneous tissue of the knee
- Femoral Nerve Block (FNB) (Active Comparator): a femoral nerve block is an anaesthetic technique that consists of anesthetizing the femoral nerve proximal of the operating area to achieve numbness distal of the block puncture site. A catheter can be placed, so the nerve can be anesthetized continuously or repeatedly for post-operative pain relieve.
  In this study the FNB with catheter will be combined with local infiltration analgesia (LIA) of the posterior capsule of the knee
  Interventions: Procedure: LIA of the posterior capsule of the knee; Procedure: FNB with catheter

INTERVENTIONS:
Procedure: LIA of the posterior capsule of the knee — the surgeon infiltrates the posterior capsule of the knee using 100 mL ropivacaine 0.2% with 0.5 mg epinephrine.
  Other Names: Naropin 0.2%; Adrenalin 1mg/mL; local infiltration analgesia
Procedure: LIA of the anterior capsule of the knee — the surgeon infiltrates the anterior capsule of the knee using 50 mL ropivacaine 0.2% with 0.25 mg epinephrine.
  Other Names: Naropin 0.2%; Adrenalin 1mg/mL; local infiltration analgesia
  Arms: Local Infiltration Analgesia (LIA)
Procedure: LIA of the subcutaneous tissue of the knee — the surgeon infiltrates the subcutaneous tissue of the knee using 50 mL ropivacaine 0.2% before wound closure.
  Other Names: Naropin 0.2%; local infiltration analgesia
  Arms: Local Infiltration Analgesia (LIA)
Procedure: FNB with catheter — pre-operatively the anesthesiologist will ultrasound guided place a catheter close to the femoral nerve using sodium chloride (NaCl 0.9%) (no local anesthetic). During surgery, when the LIA of the posterior capsule is performed, 20 mL ropivacaine 0.2% will be administered through the catheter to create a femoral nerve block (FNB). Postoperatively patients will receive 20 mL ropivacaine 0.2% through the catheter 6 times daily for 24 hours
  Other Names: Naropin 0.2%; normal saline; femoral nerve block; continuous femoral nerve block; femoral catheter
  Arms: Femoral Nerve Block (FNB)

SUMMARY:
The objective of this study is to determine whether either a femoral nerve block (FNB) or local infiltration analgesia (LIA) is a better anesthetic technique to achieve optimal functional outcome after one year in patients receiving a total knee arthroplasty and following a fast track rehabilitation protocol.

DETAILED DESCRIPTION:
For an optimal and fast recovery after total knee arthroplasty (TKA), a fast track rehabilitation protocol has been developed. The literature is not yet conclusive about the optimal anesthestic technique. The optimal technique should support fast mobilization by giving good pain relieve with minimal side effects such as nausea, drowsiness and muscle weakness. If pain relieve is optimal, the patient mobilizes fast and length of stay is shortened. But does fast recovery lead to better functional outcome? The objective of this study is to determine whether either a femoral nerve block (FNB) or local infiltration analgesia (LIA) is a better anesthetic technique to achieve optimal functional outcome after one year in patients receiving a total knee arthroplasty and following a fast track rehabilitation protocol.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical health status I-II
* patient presents with non-inflammatory primary knee osteoarthritis (radiological confirmation)
* patient is planned for a primary unilateral posterior-stabilized tri-compartmental cemented total knee replacement (Genesis II - PS)
* patient is scheduled for fast track protocol
* patient plans to be available fot follow-up through one year post-operative
* written informed consent

Exclusion Criteria:

* any contra-indication for locoregional anesthesia
* any contra-indication for spinal anesthesia
* traumatic osteoarthritis requiring TKA
* an active, local infection or systemic infection
* known hypersensitivity to amide-type local anesthetics
* known intolerance or contraindication for opioids, nonsteroidal antiinflammatory drugs (NSAIDs) or paracetamol
* a Body Mass Index > 40 kg/m2
* inability to walk independently (inability to walk at least 10 consecutive meters without a walking aid)
* scheduled for contralateral TKA within one year postoperative
* scheduled for another operation within 3 months postoperative
* physical, emotional or neurological conditions that would compromize compliance with postoperative rehabilitation and follow-up
* chronic opioid analgesic therapy
* chronic gabapentin or pregabalin analgesic therapy
* rheumatoid arthritis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rudolf Stienstra, MD, PhD, Principal Investigator — Sint Maartenskliniek
Locations (1):
- Sint Maartenskliniek, Ubbergen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fenten MGE, Bakker SMK, Scheffer GJ, Wymenga AB, Stienstra R, Heesterbeek PJC. Femoral nerve catheter vs local infiltration for analgesia in fast track total knee arthroplasty: short-term and long-term outcomes. Br J Anaesth. 2018 Oct;121(4):850-858. doi: 10.1016/j.bja.2018.05.069. Epub 2018 Jul 26. PMID 30236246

RESULTS

PARTICIPANT FLOW:
Groups:
- Femoral Nerve Block (FNB): a femoral nerve block is an anaesthetic technique that consists of anesthetizing the femoral nerve proximal of the operating area to achieve numbness distal of the block puncture site. A catheter can be placed, so the nerve can be anesthetized continuously or repeatedly for post-operative pain relieve.
  In this study the FNB with catheter will be combined with local infiltration analgesia (LIA) of the posterior capsule of the knee
  LIA of the posterior capsule of the knee: the surgeon infiltrates the posterior capsule of the knee using 100 mL ropivacaine 0.2% with 0.5 mg epinephrine.
  FNB with catheter: pre-operatively the anesthesiologist will ultrasound guided place a catheter close to the femoral nerve using sodium chloride (NaCl 0.9%) (no local anesthetic). During surgery, when the LIA of the posterior capsule is performed, 20 mL ropivacaine 0.2% will be administered through the catheter to create a femoral nerve block (FNB). Postoperatively patients will receive 20 mL ropivacaine 0.2% through the catheter 6 times daily for 24 hours
Period: Overall Study
Arm/Group | Local Infiltration Analgesia (LIA) | Femoral Nerve Block (FNB)
Started | 40 | 40
Completed | 40 | 40
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Infiltration Analgesia (LIA) | Femoral Nerve Block (FNB) | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (6.9) | 66 (6.3) | 65 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 20 | 17 | 37
Region of Enrollment [Number; unit: participants]
  Netherlands | 40 | 40 | 80
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.4 (4.2) | 30.0 (4.9) | 29.2 (4.6)
ASA physical status [Count of Participants; unit: Participants] — For full table on the ASA Physical Status Classification system and the use of examples see https://www.asahq.org/standards-and-guidelines/asa-physical-status-classification-system.
  In short: ASA 1: normal healthy patient; ASA 2 a patient with mild systemic disease; ASA 3 A patient with severe systemic disease, ASA 4 a patient with severe systemic disease that is a constant thread to life; ASA 5 a moribunt patient who is not expected to survive without the operation; ASA 6 a declared brain-dead patient whose organs are being removed for donor purposes
  Participants
    ASA 1 | 13 | 8 | 21
    ASA 2 | 15 | 24 | 39
    ASA 3 | 12 | 8 | 20
Side of surgery [Count of Participants; unit: Participants]
  left | 17 | 22 | 39
  right | 23 | 18 | 41

OUTCOME MEASURES:

1. Primary Outcome: Stair Climbing Task (SCT)
Description: The SCT assesses the ability to ascend and descend a flight of stairs, as well as lower extremity strength, power, and balance.
Time Frame: one year
Population: One patient from group FNB was excluded due to revision surgery of the knee; one patient from group FNB withdrew from follow up due to the development of a malignancy. One patient in group FNB and three patients in group LIA were excluded due to TKA of the contralateral knee. In group LIA one patient withdrew from follow up due to the development of a severe eye disorder requiring intensive treatment. One patient from group FNB was unable to perform the 6MWT due to severe backache.
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Local Infiltration Analgesia (LIA) | Femoral Nerve Block (FNB)
Number analyzed (Participants) | 36 | 37
seconds | 14.3 (7.1) | 13.8 (4.7)

2. Secondary Outcome: Timed Up and Go Test (TUG)
Description: The TUG assesses basic mobility skill as well as strength, balance, and agility. Originally developed for frail elderly people as the "Get-Up and Go Test" in 1986, it was adapted in 1991 to include the "time" component. The TUG is used in a range of populations from children to the elderly and for many conditions, including osteoarthritis, joint arthroplasty, rheumatoid arthritis, hip fractures, stroke, vertigo, and cerebral palsy.
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Local Infiltration Analgesia (LIA) | Femoral Nerve Block (FNB)
Number analyzed (Participants) | 36 | 37
seconds | 7.8 (1.9) | 7.6 (1.2)

3. Secondary Outcome: Six Minute Walking Test (6MWT)
Description: The 6MWT assesses endurance and ability to walk over longer distances. The 6MWT was first described as a field test for physical fitness in 1963 and then as a 12-minute walk test in people with chronic bronchitis. The 6MWT was found to perform as well as the 12-minute walk, and is now used to assess the submaximal level of functional performance at a similar level required for daily physical activities.
  Used in many conditions, such as osteoarthritis, cardiopulmonary disease, stroke, traumatic brain injury, patients who have undergone an amputation, Parkinson's disease, and Alzheimer's disease, as well as in elderly populations and children.
Time Frame: 1 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Local Infiltration Analgesia (LIA) | Femoral Nerve Block (FNB)
Number analyzed (Participants) | 36 | 36
meters | 489 (71) | 505 (84)

ADVERSE EVENTS:
Arm/Group | Local Infiltration Analgesia (LIA) | Femoral Nerve Block (FNB)
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 0/40 | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes